CLINICAL TRIAL: NCT00049894
Title: Predictors of Recurrent Stroke in the PROGRESS Study
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1201; R01HL071685 (NIH)
Record Dates: First submitted 2002-11-14; First posted 2002-11-15 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2005-10

CONDITIONS: Cardiovascular Diseases; Cerebrovascular Accident; Cerebrovascular Disorders; Hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Stroke; Cerebrovascular Disorders; Hypertension

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
To investigate mechanisms of recurrent stroke.

DETAILED DESCRIPTION:
BACKGROUND:

There was an urgent need to design more effective stroke prevention strategies. Previous prevention strategies including blood pressure control and anti-platelet therapy resulted in only a 43% reduction in stroke risk in a multi-center study, PROGRESS. Other proposed potentially modifiable mechanisms that mediated endothelial cell injury and activation leading to accelerated atherosclerosis including dyslipidemia, oxidative stress, endothelial dysfunction, inflammation, and renin-angiotensin system (RAS) activation were candidate strategies. Plasma markers of these various proposed mechanisms were studied to see if they predicted recurrent stroke. Since strokes kill 5 million people each year, at least one third of the 15 million others who sustain a non-fatal stroke suffer permanent disability, and those who have a transient ischemic attack (TIA) are also likely to have a recurrent event, identifying potentially modifiable risk factors would significantly reduce morbidity and mortality due to strokes worldwide.

The study was based on plasma samples taken on enrollment from a subset of the 6,105 subjects in the Perindopril Protection Against Recurrent Stroke Study (PROGRESS). The PROGRESS was an international, randomized, double-blind controlled study of a perindopril-based blood pressure lowering regimen among individuals with stroke or transient ischemic attack within the previous five years. Coordination and monitoring for PROGRESS were maintained through two international coordinating centers, one in Sydney, Australia and the other in Auckland and through seven regional coordinating centers in Beijing, Glasgow, Melbourne, Milan, Osaka, Paris and Uppsala. There were 172 local clinical centers distributed through 10 countries: Australia, Belgium, China, France, Ireland, Italy, Japan, New Zealand, Sweden and the United Kingdom.

The study was in response to a Request for Applications entitled "NHLBI Innovative Research Grant Program" released in July, 2001. The purpose of the initiative was to support new approaches to heart, lung, and blood diseases and sleep disorders that used existing data sets or existing biological specimen collections whether obtained through National Heart, Lung, and Blood Institute support or not.

DESIGN NARRATIVE:

This was a nested case-control study. Plasma samples were obtained from 6,105 subjects enrolled in the PROGRESS study, The nested case-control study included 1773 patients: 591 were cases (83 hemorrhagic strokes, 472 ischemic strokes, and 36 of unknown type), and 1182 were controls who did not subsequently become cases. Controls satisfying all matching criteria were found for 572 of these cases; 19 were incompletely matched. After the addition of cases who acted as matched controls for other cases and taking account of controls who acted for >1 case, there were 33 cases with 1, 213 with 2, and 345 with 3 matched controls. Altogether, 89 cases served as controls for 1 other case. The data were related to clinical markers of cardiovascular risk on enrollment. The study was designed to determine which of these plasma markers provided an independent measure of risk of recurrent stroke. In addition, the study determined those plasma markers that provided an independent measure of reduction in risk of recurrent stroke by perindopril-based antihypertensive therapy, thereby providing a means to identify those subjects most likely to benefit from such therapy, and conversely, those subjects in whom alternative preventative strategies were required. In addition, plasma markers that predicted risk of recurrent stroke may have indicated novel therapies to prevent this condition.

Specific aims included identifying whether nuclear magnetic resonance-determined lipoprotein profiles, and plasma levels of homocysteine, protein carbonyls, chlorotyrosine, soluble vascular cell adhesion molecule (sVCAM-1), C-reactive peptide (CRP), active renin, and the amino-terminal pro-B-type natriuretic peptide (NT-proBNP) predicted recurrent stroke in PROGRESS study participants and whether these measures predicted benefit from perindopril-based antihypertensive therapy.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2002-09; Study Completion 2004-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Duncan Campbell — St Vincent's Institute of Medical Research

REFERENCES:
- [Background] Campbell DJ, Woodward M, Chalmers JP, Colman SA, Jenkins AJ, Kemp BE, Neal BC, Patel A, MacMahon SW. Prediction of heart failure by amino terminal-pro-B-type natriuretic peptide and C-reactive protein in subjects with cerebrovascular disease. Hypertension. 2005 Jan;45(1):69-74. doi: 10.1161/01.HYP.0000151103.02424.c3. Epub 2004 Nov 29. PMID 15569851
- [Background] Woodward M, Lowe GD, Campbell DJ, Colman S, Rumley A, Chalmers J, Neal BC, Patel A, Jenkins AJ, Kemp BE, MacMahon SW. Associations of inflammatory and hemostatic variables with the risk of recurrent stroke. Stroke. 2005 Oct;36(10):2143-7. doi: 10.1161/01.STR.0000181754.38408.4c. Epub 2005 Sep 8. PMID 16151030